CLINICAL TRIAL: NCT02765516
Title: Genetic Basis for Prediction of Non-responders to Dietary Plant Sterol Intervention
Acronym: GenePredict-PS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit
Sponsor: University of Manitoba (Other)
Collaborators: Mitacs (Industry); Unilever R&D (Industry); Nutritional Fundamentals for Health (Unknown)
Responsible Party: Principal Investigator, Dr. J. House, Head/Professor, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: MITACS Converge MC00009
Record Dates: First submitted 2016-04-22; First posted 2016-05-06 (Estimated); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Hypercholesterolemia; Cardiovascular Disease
MeSH Terms: conditions — Hypercholesterolemia; Cardiovascular Diseases | interventions — Phytosterols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant sterols (Active Comparator)
  Interventions: Other: Plant sterols
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Plant sterols — 2.0g/day of plant sterols incorporated into margarine to be consumed for 28 days
  Arms: Plant sterols
Other: Placebo — Identical margarine without additional plant sterols to be consumed for 28 days
  Arms: Placebo

SUMMARY:
The objective of this study is to utilize information on associations between genetic predisposition pertaining to multiple single nucleotide polymorphisms (SNPs) and the degree of responsiveness of low-density lipoprotein cholesterol (LDL-C) lowering to plant sterols (PS). The predictive potential of SNPs associated with PS responsiveness will be evaluated using a randomized human intervention trial examining responsiveness of lowering blood LDL-C levels to PS intervention.

DETAILED DESCRIPTION:
On average plant sterol (PS) consumption of 2-3 grams a day leads to a ~10% decrease in low-density lipoprotein cholesterol (LDL-C). However, inter-individual response to PS consumption varies, with some individuals showing low or no reductions in LDL-C levels, while some even showing an increase in levels. Determining factors that predict the direction of response of LDL-C to PS would be helpful in identifying individuals who should consume PS and individuals who should seek another method of treating hypercholesterolemia. The objective of this research proposal is to test the a priori predictive potential of a combination of three single nucleotide polymorphisms (SNPs), i.e., genosets, previously associated with response to PS in a post-hoc manner. A clinical trial with a priori recruitment of participants based on genoset which will test LDL-C response to PS consumption using a randomized, double blind, placebo controlled crossover design is proposed.

ELIGIBILITY:
Inclusion Criteria:

* Fasting LDL-C concentration >3.0 and <4.9 mmol/L
* Fasting glucose concentration <6.1 mmol/L
* Fasting triglyceride concentration <4.52 mmol/L
* Genoset required: ; ApoE ε3/ε3 CYP7A1 rs3808607 T/T (n=20); ApoE ε3/ε3 CYP7A1 rs3808607 G/- (n=22); ApoE ε4/- CYP7A1 rs3808607 -/- (n=22)

Exclusion Criteria:

* Consuming, or have consumed in the last 3 months, medications or nutritional supplements which are known to affect lipid metabolism (such as cholestyramine, colestipol, niacin, clofibrate, gemfibrozil, probucol, HMG-CoA R inhibitors, methotrexate, high dose dietary supplements, fish oil capsules or plant sterol or stanol), or have any dietary restrictions which would prevent them from consuming the trial treatments
* BMI >40
* Must not have self-reported weight gain or loss greater than 3 kg in the past three months
* Phytosterolemic
* History of active cardiovascular disease including stroke, congestive heart failure, myocardial infarction, unstable angina pectoris, coronary artery bypass graft, percutaneous transluminal coronary angioplasty, temporal ischemic attacks, anemia, abnormal electrolytes, proteinuria, and abnormal liver, kidney or thyroid function
* Type 1 or type 2 diabetes, a history of cancer or malignancy in the last 5 years, or any metabolic disease, gastrointestinal disorder or other clinically significant disease/disorder which could interfere with the results of the study or the safety of the participant.
* Uncontrolled hypertension having systolic blood pressure >160mm Hg or diastolic blood pressure >100mm Hg
* Smoker, tobacco/snuff/nicotine users, recreational drug users
* Consume more than 14 alcoholic beverages a week
* Participants who are pregnant or plan to become pregnant during the trial period or lactating mothers
* Participants will be excluded if they have clinically significant biochemistry defined as: LDL-C <3.0mmol/L or >4.9 mmol/L; TC > 6.2 mmol/L; fasting glucose: > 6.1 mmol/ l, fasting TG >4.52 mmol/L; AST >100 U/L; ALT >100 U/L or or any other clinically significant abnormality in hematology and/or biochemistry at the investigator's discretion
* Patients with unstable or serious illness, for example, dementia, terminal illness, recent bereavement, recent significant medical diagnosis will also be excluded

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in fasting low-density lipoprotein cholesterol (LDL-C) levels between placebo and treatment endpoints (in a crossover design) | Endpoint (Days 28,29) of each treatment period

SECONDARY OUTCOMES:
Change in fasting total cholesterol (TC) levels between placebo and treatment endpoints (in a crossover design) | Endpoint (Days 28,29) of each treatment period
Change in fasting high-density lipoprotein cholesterol levels between placebo and treatment endpoints | Endpoint (Days 28,29) of each treatment period
Change in fasting triglyceride (TG) levels between placebo and treatment endpoints (in a crossover design) | Endpoint (Days 28,29) of each treatment period
Change in body weight between placebo and treatment endpoints (in a crossover design) | Endpoint (Days 28,29) of each treatment period
Change in body mass index (BMI) between placebo and treatment endpoints (in a crossover design) | Endpoint (Days 28,29) of each treatment period
Change in waist circumference between placebo and treatment endpoints (in a crossover design) | Endpoint (Days 28,29) of each treatment period
Change in blood pressure between placebo and treatment endpoints (in a crossover design) | Endpoint (Days 28,29) of each treatment period
Change in arterial stiffness-Pulse wave velocity between placebo and treatment endpoints (in a crossover design) | Endpoint (Days 28,29) of each treatment period
  Pulse wave velocity will be determined using an automated oscillometric measurement device (Mobil-O-Graph, IEM, Stolberg, Germany).
Change in arterial stiffness-augmentation index between placebo and treatment endpoints (in a crossover design) | Endpoint (Days 28,29) of each treatment period
  Augmentation index will be determined using an automated oscillometric measurement device (Mobil-O-Graph, IEM, Stolberg, Germany).
Change in fasting glucose levels between placebo and treatment endpoints (in a crossover design) | Endpoint (Days 28,29) of each treatment period
Change in blood sterols and sterol precursors (non-cholesterol sterols) levels between placebo and treatment endpoints (in a crossover design) | Endpoint (Days 28,29) of each treatment period
Change in fractional cholesterol synthesis between placebo and treatment endpoints (in a crossover design) | Endpoint (Day 28,29) of each treatment period
  A fasted blood sample will be taken on day 28 of each study period prior to deuterium oxide administration, as well as fasting samples on day 29. The change in deuterium enrichment within red blood cell (RBC) free cholesterol we be determined as an index of synthesis over days 28 and 29.

CONTACTS AND LOCATIONS:
Overall Officials: James House, PhD, Principal Investigator — University of Manitoba; Dylan Mackay, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Department of Human Nutritional sciences, University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shamloo M, Granger MJ, Trautwein EA, House JD, MacKay D. Genetic basis for prediction of non-responders to dietary plant sterol intervention (GenePredict-PS): a study protocol for a double-blind, placebo-controlled, randomized two-period crossover study. Trials. 2020 Jun 1;21(1):452. doi: 10.1186/s13063-020-04364-5. PMID 32487131